CLINICAL TRIAL: NCT05101603
Title: Effects of Nd:YAG Laser and Air Abrasive Combined Application on Clinical Parameters in Addition to Non Surgical Periodontal Treatment in Patients With Periodontitis
Brief Title: Effects of Nd:YAG Laser and Air Abrasive Combined Application in Patients With Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, İsmet İlke ALKAN, Research Assistant Dentist, Izmir Katip Celebi University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: IsmetIlke
Record Dates: First submitted 2021-10-07; First posted 2021-11-01 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Periodontitis
Keywords: Periodontitis; Non surgical periodontal treatment; Nd:YAG laser; Perioflow; Erythritol Powder
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Only non surgical periodontal treatment
  Interventions: Procedure: Non surgical periodontal therapy
- Test (Experimental): Nd:YAG Laser and air abrasive combined application addition to non surgical periodontal treatment
  Interventions: Device: Air Abrasive; Device: Nd:YAG Laser; Procedure: Non surgical periodontal therapy

INTERVENTIONS:
Device: Air Abrasive — Applied with Nd:YAG Laser on periodontal pockets
  Other Names: EMS Dental Air-Flow® Handy Perio, Switzerland
  Arms: Test
Device: Nd:YAG Laser — Applied with Air Abrasive on periodontal pockets
  Other Names: Fotona Fidelis AT, Ljubljana, SLOVENIA
  Arms: Test
Procedure: Non surgical periodontal therapy — The first phase, in which optimum plaque control is achieved and local etiological factors are removed, is the first step of all periodontal diseases and surgical procedures.

SUMMARY:
The aim of this clinical study is to investigate the effectiveness of the combined application of Nd:YAG (neodymium-doped yttrium aluminum garnet) laser and air abrasive applied in addition to nonsurgical periodontal treatment on clinical parameters in patients with periodontitis.

A split-mouth, randomized study included 24 systemically healthy, non-smoker, periodontitis patients. In addition to non-surgical periodontal treatment, air abrasive (erythritol-chlorhexidine powder) and Nd:YAG laser (2 W, 200mJ, 10 Hz) combined application was applied to the test group, while only non-surgical periodontal treatment was applied to the control group. Clinical periodontal records of the patients, including plaque index (PI), gingival index (GI), bleeding on probing (BOP), probing pocket depth (PD), clinical attachment level (CAL), were taken before the treatment and at the 1st and 3rd months after the treatment.

All clinical parameters improved significantly from baseline for both groups after treatment (p˂0.05). In the evaluation between the test and control groups, no statistically significant difference was found in the PI, GI and BOP parameters of the patients at any time (p˃0.05). While the amount of change in PD and CAL values after treatment in medium deep pockets in the study groups was compared, no significant difference was observed between the groups (p˃0.05), statistically significant improvements in PD and CAL parameters were observed in the test group compared to the control group only for deep pockets (≥7 mm) among the groups (p˂0.05).In conclusion, it has been observed that the combined application of Nd:YAG laser and air abrasive in systemically healthy, stage III and grade C periodontitis patients is in the short term on PD and CAL, especially in inaccessible areas such as deep pockets.

DETAILED DESCRIPTION:
Recently, erythritol has been introduced as a new air abrasive powder. Erythritol is a sugar alcohol. It is a water-soluble, chemically neutral artificial sweetener. Compared to glycine, another powder used in air abrasive devices, erythritol has a smaller particle size. Subgingival air abrasive application with erythritol has been shown to effectively remove subgingival biofilm from the root surface. In addition, erythritol has been reported to suppress bi-species biofilm formation of Porphyromonas gingivalis (p. gingivalis) and Streptococcus gordonii (s. gordonii) through ribonucleic acid (RNA) and deoxyribonucleic acid (DNA) depletion and metabolic changes.

In recent years, lasers have gained increasing interest in the treatment of periodontitis as an adjunct or alternative treatment procedure to conventional treatment. It has been stated that the Nd:YAG laser provides excellent tissue ablation with strong bactericidal and detoxification effects, and it has been shown that it can reach deep pockets that conventional instruments cannot reach (7,19). It has been reported that Nd:YAG laser creates a very thick coagulation layer on soft tissue surfaces. It has also been proven that when applied to the pockets, it can remove the infected pocket epithelium. When applied in addition to non-surgical periodontal therapy, it has been shown to dramatically improve the clinical manifestations of periodontal inflammation compared to conventional therapy.

In this clinical study, it was aimed to clinically evaluate the effectiveness of subgingival Nd:YAG laser and air abrasive combined application in addition to non-surgical periodontal treatment in systemically healthy periodontitis patients. The efficacy of the combined Nd:YAG laser and air abrasive application was evaluated by examining the clinical periodontal parameters of the patients [plaque index (PI), probing pocket depth (PD), gingival index (GI), probing bleeding index (BI) and clinical attachment level (CAL)].

It is thought that, in addition to non-surgical periodontal treatment, YAG laser and air abrasive combined applications will have an antimicrobial effect on the biofilm in difficult areas and deep pockets that hand tools cannot reach, provide better penetration than irrigation fluids and contribute to periodontal regeneration. Thus, it is hoped to increase clinical success, prevent disease recurrences, reduce the need for periodontal surgery and increase the quality of life of patients.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy (The determination of healthy volunteers will be based on the statements of the patients in the anamnesis. No additional examinations will be made.),
* Having a total of at least twenty permanent teeth in the mouth,
* Non-smoker
* Have not used antibiotics, anti-inflammatory and systemic corticosteroid drugs in the last 6 months,
* Not in pregnancy or lactation period,
* Patients who have not received periodontal treatment in the last 6 months,
* Patients who accepted the research and signed the informed volunteer consent form
* Bleeding on probing in 30% or more areas,
* 5 mm or more probing pocket depth in each quadrant in at least 2 non-adjacent teeth
* 4mm or more attachment loss,
* Coronal 1/3 or more (horizontal and/or vertical) on radiograph individuals with bone loss were included

Exclusion Criteria:

* Having any systemic disease,
* Regularly using a systemic medication,
* Being pregnant or lactating.
* To have had periodontal treatment in the last 6 months.
* Receiving antibiotic, anti-inflammatory or systemic corticosteroid medication in the last 6 months.
* Smoking.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Clinical attachment level change | Change from baseline clinical attachment level at 3 months
  With the help of a Williams periodontal probe, the distance between the enamel-cementum border and the sulcus/pocket floor will be measured from the six points of the tooth: mesiobuccal, midbuccal, distobuccal, mesiopalatal/lingual, mid-buccal/palatal and distobuccal/palatal.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Sağlam, Study Director — Izmir Katip Celebi University Faculty of Dentistry
Locations (1):
- Izmir Katip Celebi University Faculty of Dentistry, Izmir, Çiğli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hagi TT, Hofmanner P, Salvi GE, Ramseier CA, Sculean A. Clinical outcomes following subgingival application of a novel erythritol powder by means of air polishing in supportive periodontal therapy: a randomized, controlled clinical study. Quintessence Int. 2013 Nov-Dec;44(10):753-61. doi: 10.3290/j.qi.a30606. PMID 24078975
- [Background] Hashino E, Kuboniwa M, Alghamdi SA, Yamaguchi M, Yamamoto R, Cho H, Amano A. Erythritol alters microstructure and metabolomic profiles of biofilm composed of Streptococcus gordonii and Porphyromonas gingivalis. Mol Oral Microbiol. 2013 Dec;28(6):435-51. doi: 10.1111/omi.12037. Epub 2013 Jul 29. PMID 23890177
- [Background] Crespi R, Covani U, Margarone JE, Andreana S. Periodontal tissue regeneration in beagle dogs after laser therapy. Lasers Surg Med. 1997;21(4):395-402. doi: 10.1002/(sici)1096-9101(1997)21:43.0.co;2-a. PMID 9328987
- [Background] Ting CC, Fukuda M, Watanabe T, Sanaoka A, Mitani A, Noguchi T. Morphological alterations of periodontal pocket epithelium following Nd:YAG laser irradiation. Photomed Laser Surg. 2014 Dec;32(12):649-57. doi: 10.1089/pho.2014.3793. PMID 25392971
- [Background] Gold SI, Vilardi MA. Pulsed laser beam effects on gingiva. J Clin Periodontol. 1994 Jul;21(6):391-6. doi: 10.1111/j.1600-051x.1994.tb00735.x. PMID 8089240
- [Background] Qadri T, Poddani P, Javed F, Tuner J, Gustafsson A. A short-term evaluation of Nd:YAG laser as an adjunct to scaling and root planing in the treatment of periodontal inflammation. J Periodontol. 2010 Aug;81(8):1161-6. doi: 10.1902/jop.2010.090700. PMID 20397904
- [Background] Nagy RJ, Otomo-Corgel J, Stambaugh R. The effectiveness of scaling and root planing with curets designed for deep pockets. J Periodontol. 1992 Dec;63(12):954-9. doi: 10.1902/jop.1992.63.12.954. PMID 1474467
- [Background] Papapanou PN, Sanz M, Buduneli N, Dietrich T, Feres M, Fine DH, Flemmig TF, Garcia R, Giannobile WV, Graziani F, Greenwell H, Herrera D, Kao RT, Kebschull M, Kinane DF, Kirkwood KL, Kocher T, Kornman KS, Kumar PS, Loos BG, Machtei E, Meng H, Mombelli A, Needleman I, Offenbacher S, Seymour GJ, Teles R, Tonetti MS. Periodontitis: Consensus report of workgroup 2 of the 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions. J Clin Periodontol. 2018 Jun;45 Suppl 20:S162-S170. doi: 10.1111/jcpe.12946. PMID 29926490
- [Background] Badersten A, Nilveus R, Egelberg J. Effect of nonsurgical periodontal therapy. II. Severely advanced periodontitis. J Clin Periodontol. 1984 Jan;11(1):63-76. doi: 10.1111/j.1600-051x.1984.tb01309.x. PMID 6363463
- [Background] Drisko CH. Nonsurgical periodontal therapy. Periodontol 2000. 2001;25:77-88. doi: 10.1034/j.1600-0757.2001.22250106.x. PMID 11155183
- [Background] Petersilka GJ, Bell M, Mehl A, Hickel R, Flemmig TF. Root defects following air polishing. J Clin Periodontol. 2003 Feb;30(2):165-70. doi: 10.1034/j.1600-051x.2003.300204.x. PMID 12622860
- [Background] Petersilka G. Re: "Subgingival plaque removal using a new air-polishing device". Moene R, Decaillet F, Andersen E, Mombelli A. (J Periodontol 2010;81:79-88.). J Periodontol. 2010 Jul;81(7):962-3. doi: 10.1902/jop.2010.100118. No abstract available. PMID 20553116
- [Background] Cobb CM, Daubert DM, Davis K, Deming J, Flemmig TF, Pattison A, Roulet JF, Stambaugh RV. Consensus Conference Findings on Supragingival and Subgingival Air Polishing. Compend Contin Educ Dent. 2017 Feb;38(2):e1-e4. PMID 28156118
- [Background] Munro IC, Berndt WO, Borzelleca JF, Flamm G, Lynch BS, Kennepohl E, Bar EA, Modderman J. Erythritol: an interpretive summary of biochemical, metabolic, toxicological and clinical data. Food Chem Toxicol. 1998 Dec;36(12):1139-74. doi: 10.1016/s0278-6915(98)00091-x. PMID 9862657